CLINICAL TRIAL: NCT01736865
Title: Vitamin D for Established Type 2 Diabetes (DDM2)
Acronym: DDM2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK76092-06; R01DK076092 (NIH)
Record Dates: First submitted 2012-11-15; First posted 2012-11-29 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): One placebo pill daily for 1 year
  Interventions: Drug: Placebo
- cholecalciferol (Active Comparator): One cholecalciferol pill daily for 1 year
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol
  Arms: cholecalciferol
Drug: Placebo
  Arms: placebo

SUMMARY:
This research study in adults with established type 2 diabetes will test whether daily vitamin D supplementation affects how the body processes glucose (sugar).

ELIGIBILITY:
Inclusion Criteria:

* Established type 2 diabetes, defined by one of the following two criteria:
* Age ≥ 25 years and ≤ 75 years
* BMI: 23 to 40 kg/m2 inclusive
* Provision of signed and dated written informed consent prior to any study procedures.

Major Exclusion Criteria

* "Severe" diabetes defined by one of the following criteria:
* - (a) Symptoms of hyperglycemia;
* - (b) Screening HbA1c ≥ 7.5 [may indicate potential for rapid progression during the trial necessitating need to amplify diabetes-specific pharmacotherapy]
* History of nephrolithiasis or hypercalcemia

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2012-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Cincinnati VA Medical Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Meng H, Matthan NR, Angellotti E, Pittas AG, Lichtenstein AH. Exploring the effect of vitamin D3 supplementation on surrogate biomarkers of cholesterol absorption and endogenous synthesis in patients with type 2 diabetes-randomized controlled trial. Am J Clin Nutr. 2020 Sep 1;112(3):538-547. doi: 10.1093/ajcn/nqaa149. PMID 32559272
- [Derived] Angellotti E, D'Alessio D, Dawson-Hughes B, Chu Y, Nelson J, Hu P, Cohen RM, Pittas AG. Effect of vitamin D supplementation on cardiovascular risk in type 2 diabetes. Clin Nutr. 2019 Oct;38(5):2449-2453. doi: 10.1016/j.clnu.2018.10.003. Epub 2018 Oct 9. PMID 30352748
- [Derived] Alzaman NS, Dawson-Hughes B, Nelson J, D'Alessio D, Pittas AG. Vitamin D status of black and white Americans and changes in vitamin D metabolites after varied doses of vitamin D supplementation. Am J Clin Nutr. 2016 Jul;104(1):205-14. doi: 10.3945/ajcn.115.129478. Epub 2016 May 18. PMID 27194308

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 127 participants were enrolled because by the time the 124 "needed" was reached, 3 additional participants were eligible and wanted to be part of the trial.
Groups:
- Placebo: One placebo pill daily for 1 year
  Placebo
- Cholecalciferol: One cholecalciferol pill daily for 1 year
  Cholecalciferol
Period: Overall Study
Arm/Group | Placebo | Cholecalciferol
Started | 61 | 66
Completed | 61 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cholecalciferol | Total
Number analyzed (Participants) | 61 | 66 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.5) | 60.1 (8.4) | 60.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 40 | 49 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 60 | 60 | 120
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 17 | 38
  White | 38 | 41 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/ m2] | 31.2 (3.8) | 30.7 (3.9) | 30.9 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Disposition Index
Description: Disposition index by the insulin secretion sensitivity index-2 (ISSI-2). This is an calculated value which represents the ability of a person's pancreatic beta cells to lower blood glucose. A higher number means the pancreas is better able to secrete insulin and improve glucose levels.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: index
Arm/Group | Placebo | Cholecalciferol
Number analyzed (Participants) | 59 | 61
index | 0.023 (0.057) | 0.149 (0.056)

2. Secondary Outcome: Number of Participants With Change in Glycemia
Description: Change in glycemia (categorical variable, composite outcome) defined as [1] a decrease in diabetes medications or [2] a reduction of equal to or more than 0.4 HbA1c units from baseline without increasing medications.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cholecalciferol
Number analyzed (Participants) | 59 | 61
Participants | 53 | 52

3. Other Pre Specified Outcome: Hemoglobin A1c
Time Frame: 12 months
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Placebo | Cholecalciferol
Number analyzed (Participants) | 59 | 61
percentage | 0.2 (0.07) | 0.2 (0.06)

4. Other Pre Specified Outcome: Change in Diabetes Medications
Time Frame: 6 and 12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Variability of Response to Vitamin D Supplementation in Subgroups.
Description: Variability of response to vitamin D supplementation in subgroups defined by baseline characteristics: (1) race; (3) 25OHD concentration; (3) diabetes treatment.
Time Frame: Baseline and 12 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Effect of Vitamin D Supplementation on Blood 25-hydroxyvitaminD Concentration
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Cholecalciferol
Number analyzed (Participants) | 61 | 66
ng/mL | 27.5 (12.0) | 25.8 (10.3)

7. Other Pre Specified Outcome: Cardiovascular Risk Factors
Description: Cardiovascular risk factors defined as blood pressure, lipid profile, C-reactive protein and urine albumin excretion
Time Frame: 6 and 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Effect of Vitamin D Supplementation on Plasma Concentrations of Surrogate Biomarkers of Cholesterol Absorption (Campesterol and β-sitosterol) and Endogenous Synthesis (Lathosterol and Desmosterol)
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Placebo | Cholecalciferol
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/66
Serious Adverse Events (participants affected / at risk) | 6/61 | 7/66
Other Adverse Events (participants affected / at risk) | 24/61 | 17/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=61) | Cholecalciferol (N=66)
New or prolonged hospitalization (General disorders) | 6 (6) | 7 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=61) | Cholecalciferol (N=66)
Adverse Event (General disorders) | 24 (24) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No